CLINICAL TRIAL: NCT00859118
Title: Pharmacodynamic Study of Axitinib in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO 08905; H-2008-0202 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2011-00744 (Registry Identifier: NCI Trial ID); NCT00839215 (obsolete NCT alias)
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2014-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schedule A Cohort 1 (Experimental): Axitinib 5 mg PO BID x ~2 weeks (12-14 days), followed by 1 week drug break (for cycle 1 only). After Scan#3 obtained, patients will commence with Axitinib 5 mg PO BID continuously without breaks, repeated in 3 week cycles.
  Scan#1: Baseline (days -3 to 0) Scan#2: Week 2 (between days 12-14) Scan#3: Week 3 (7 days after axitinib held) Up to 10 patients will receive 2 DCE-CT scans at week 2 and 3, coinciding with the FLT-PET scans.
  Interventions: Drug: AG-013736
- Schedule A: Cohort 2 (Experimental): Axitinib 5 mg PO BID x ~2 weeks (12-14 days), followed by 1 week drug break (for cycle 1 only). After Scan#3 obtained, patients will commence with Axitinib 5 mg PO BID continuously without breaks, repeated in 3 week cycles.
  Scan#1: Week 2 (between days 12-14) Scan#2: Week 3 (2 days after axitinib held) Scan#3: Week 3 (7 days after axitinib held) Up to 10 patients will receive 2 DCE-CT scans at week 2 and 3, coinciding with the FLT-PET scans.
  Interventions: Drug: AG-013736

INTERVENTIONS:
Drug: AG-013736 — Axitinib 5 mg PO BID x ~2 weeks (12-14 days), followed by 1 week drug break (for cycle 1 only)
  Other Names: Axitinib
  Arms: Schedule A Cohort 1
Drug: AG-013736 — Axitinib 5 mg PO BID x ~2 weeks (12-14 days), followed by 1 week drug break (for cycle 1 only). After Scan#3 obtained, patients will commence with Axitinib 5 mg PO BID continuously without breaks, repeated in 3 week cycles.
  Other Names: Axitinib
  Arms: Schedule A: Cohort 2

SUMMARY:
The main purpose of this study is to see what changes happen to the tumors while taking the axitinib and after it is stopped (during the scheduled breaks), and what changes in the tumor may be responsible for this growth. This will be done by using a special kind of scan called an 18F-FLT PET/CT.

In addition, the investigators want to find out how the drugs are processed and distributed in the human body. The investigators will also look at how different types of cancer are affected by axitinib. The investigators will also correlate vasculature kinetics extracted from the dynamic FLT PET/CT imaging with the vasculature kinetics extracted from DCE-CT.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed solid malignancy (excluding lymphoma) that is metastatic or unresectable and for which no standard therapy exists (although all solid malignancies will be enrolled, a subset will be designated for NSCL cancer will be given due to planned trials in this disease.

  * must have measurable disease
  * Must be greater than or equal to 18 years old.
  * Life expectancy of greater than 12 weeks.
  * ECOG performance status less than or equal to 2.
  * Patients must have normal organ and marrow function
  * Must be willing to undergo planned pharmacodynamic assessments, including serial PET imaging, plasma markers, and pharmacokinetic sampling.
  * Women of childbearing potential and men must use adequate form of birth (hormonal or barrier method of birth control
  * must have ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Must not havehad chemotherapy, radiotherapy, experimental therapy or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered (to grade less than or equal to 1 or baseline) from clinically significant adverse events due to agents administered more than 4 weeks earlier (alopecia and fatigue excluded).

  * Patients may not be receiving any other investigational agents.
  * Prior anti-VEGF directed therapy may be allowed only if approved by the PI
  * Must not have history of allergic reactions attributed to compounds of similar chemical or biologic composition to axitinib.
  * Must not have poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher)
* Must not require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis.

  * Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain axitinib tablets are excluded.
  * Patients with any of the following conditions are excluded:

    * Serious or non-healing wound, ulcer, or bone fracture.
    * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment.
    * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry.
    * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry.
    * History of pulmonary embolism within the past 12 months.
    * Class III or IV heart failure as defined by the NYHA functional classification system.
  * Patients without appropriate lesion on CT scan for FLT-PET/CT imaging will be excluded.
  * The eligibility of patients taking medications that are potent inducers or inhibitors of that enzyme will be determined following a review of their case by the Principal Investigator.
  * Steroid use is not recommended during axitinib treatment unless absolutely necessary
  * Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible. Patients with a history of hypothyroidism are eligible provided they are currently euthyroid.
  * Must not have known brain metastases are excluded.
  * Must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements
  * Must not be pregnant or breastfeeding.
  * Must not be HIV-positive on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2013-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine pharmacodynamic change using FLT-PET/CT scans at baseline, during axitinib exposure and washout | 1 year
To evaluate objective response of axitinib in patients with advanced solid malignancies. | 1 year

SECONDARY OUTCOMES:
To measure change in plasma VEGF levels, during axitinib exposure and withdrawal | 1 year
Correlate axitinib pharmacokinetics with response, unexpected toxicity, VEGF levels, and FLT-PET/CT change. | 1 year
Correlate vasculature kinetics extracted from the dynamic FLT PET/CT imaging with the vasculature kinetics extracted from DCE-CT | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu